CLINICAL TRIAL: NCT05880420
Title: EXPERIMENTAL STUDY A.R.C.O. (CANCER CAREGIVER REMOTE ASSISTANCE) TELEASSISTED HOME DRESSING VS/ OUTPATIENT DRESSING OF PICC CENTRAL VENOUS CATHETER (PERIPHERAL INSERTION CENTRAL VENOUS CATHETER)
Brief Title: EXPERIMENTAL STUDY A.R.C.O. (CANCER CAREGIVER REMOTE ASSISTANCE)TELEHEALTH HOME MEDICATION VS/OUTPATIENT MEDICATION OF CENTRAL VENOUS CATHETER PICC (PERIPHERALLY INSERTED CENTRAL VENOUS CATHETER)
Acronym: ARCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RS1518/21
Record Dates: First submitted 2023-03-28; First posted 2023-05-30 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - home group (Experimental)
  Interventions: Device: Caregiver operations with medication accessories
- Arm 2 - outpatient calibration (Active Comparator)
  Interventions: Device: Nurse operations with medication accessories

INTERVENTIONS:
Device: Caregiver operations with medication accessories — After at least an initial outpatient medication (24/72 hours), home medication every 7 days (caregiver) for a total of 10 weeks.
  Arms: Arm 1 - home group
Device: Nurse operations with medication accessories — Outpatient medication every week (for a total of 10 weeks). Patients adhering to this arm will be followed at the IGAV nursing clinic of the IFOs.
  Arms: Arm 2 - outpatient calibration

SUMMARY:
Cancer patients need central venous access according to the different types of chemotherapy and support drugs for their treatment path. The presence of a central vascular access brings mechanical issues, thrombotic and infectious complications that can undermine the patient's health and the life of the catheter, therefore the management of venous accesses is clinically relevant. The prevention of infections remains mainly based on correct hand washing and compliance with aseptic techniques. This is a multicenter intervention study is composed by a single experimental arm (home) and a calibration arm (outpatient). The study is designed to evaluate that the complication rate recorded in the two groups are similar.

ELIGIBILITY:
* Share patient choice
* availability at the patient's home at least once a week
* availability during on line appointment time with the tutor/video

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Acceptability | 10 weeks
  To compare the incidence of complications found in peripherally inserted central venous catheter (PICC) management in outpatient (calibration arm) vs home management to test the hypothesis that the incidence of catheter-related complications in the home management group is not higher than that observed in the outpatient group.

CONTACTS AND LOCATIONS:
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy

REFERENCES:
- [Derived] Basili P, Farina I, Terrenato I, Centini J, Volpe N, Rizzo V, Agoglia L, Paterniani A, Aprea P, Calignano P, Petrone F, Ciliberto G. Remote Assisted Home Dressing vs. Outpatient Medication of Central Venous Catheter (Peripherally Inserted Central Venous Catheter): Clinical Trial A.R.C.O. (Remote Assistance Oncology Caregiver). Nurs Rep. 2024 Jun 11;14(2):1468-1476. doi: 10.3390/nursrep14020110. PMID 38921720